CLINICAL TRIAL: NCT03084536
Title: PECS Block vs. Multimodal Analgesia for Prevention of Persistent Postoperative Pain in Breast Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201703053
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Breast Cancer Female; Cancer of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine; Gabapentin; Celecoxib; Acetaminophen; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative PECS blocks (Active Comparator): * PECS I & II block will be administered preoperatively
  * For unilateral surgeries, a PECS I block will be performed with 0.15mL/kg of 0.375% bupivacaine (maximum 10mL). The PECS II block will be performed with 0.3 mL/kg of the same solution (maximum 20mL). If there is a contralateral surgery (simple mastectomy) a PECS II block will also be performed on the other side with 0.2mL/kg of 0.375% bupivacaine (maximum 20mL)
  * To ensure blind integrity, study drug syringes will be marked only "study drug" and subject number
  * Perioperative analgesic will be encouraged.. Gabapentin 300mg, celecoxib 200mg and acetaminophen 1000mg will be administered to all patients following arrival to the preoperative area. All patients will receive premedication of 1-2 mg midazolam IV (age < 65) and 50-100 μg fentanyl IV prior to the block placement or entry to the operating room at the discretion of the regional team or operating room anesthesiologist
  Interventions: Drug: Bupivacaine; Drug: Gabapentin; Drug: Celecoxib; Drug: Acetaminophen; Drug: Midazolam; Drug: Fentanyl
- Placebo PECS blocks (Placebo Comparator): * A sham block (normal saline) will be placed preoperatively
  * To ensure blind integrity, study drug syringes will be marked only "study drug" and subject number.
  * Perioperative analgesic regimen will be encouraged. Gabapentin 300mg, celecoxib 200mg and acetaminophen 1000mg will be administered to all patients following arrival to the preoperative holding area. On the day of surgery all patients will receive premedication of 1-2 mg midazolam IV (age < 65) and 50-100 μg fentanyl IV prior to the block placement or entry to the operating room at the discretion of the regional team or operating room anesthesiologist.
  Interventions: Drug: Gabapentin; Drug: Celecoxib; Drug: Acetaminophen; Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine — -Given after general anesthesia
  Other Names: Bupivacaine hydrochloride
  Arms: Preoperative PECS blocks
Drug: Gabapentin — * As per routine care
  * Will not be prescribed for any patient with preexisting kidney disease or ≥ 65 years.
Drug: Celecoxib — * As per routine care
  * Will not be prescribed for any patient with preexisting kidney disease or ≥ 65 years.
  * Naproxen will be substituted for celecoxib in patients with sulfa allergies.
Drug: Acetaminophen — -As per routine care
Drug: Midazolam — -As per routine care
Drug: Fentanyl — -As per routine care

SUMMARY:
In this double blinded randomized placebo-controlled trial, 160 subjects scheduled for breast surgery involving the axilla will be administered a multimodal pain regimen including acetaminophen, dexamethasone, celecoxib, and gabapentin. 80 subjects will also receive a Pectoral Nerve blocks I and II (PECS I and II block) preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective breast cancer surgeries at Barnes-Jewish Hospital:

  * unilateral axillary dissection
  * unilateral modified radical mastectomy
  * mastectomy with same day unilateral reconstruction
  * unilateral sentinel lymph node biopsy (SLNB)
  * partial mastectomy with unilateral SLNB
  * simple mastectomy with unilateral SLNB
* At least 18 years of age.
* Able to understand and willing to sign an Institutional Review Board (IRB)-approved written informed consent document.
* Enrollment in the SATISFY-SOS study (WUSTL IRB# 201203088, NCT02032030).

Exclusion Criteria:

* Planned for bilateral axillary or bilateral reconstruction surgery.
* Previous surgery on the surgical breast and/or axilla with the exception of partial mastectomy or sentinel lymph node biopsy
* Pre-existing pain in the axilla affecting the ability to use extremity for activities of daily living or requiring medication for treatment.
* Current or past medical history of liver disease or cirrhosis with an elevated INR >1.4 or currently elevated transaminase levels.
* Known contraindications to peripheral nerve block placement.
* Pregnant or breastfeeding.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition
* Planned additional surgery to the surgical breast or axilla in the next year (exception would be minor surgery to breast but not axilla such as simple tissue expander replacement or lumpectomy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Guffey, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized to an Arm: -Participants were removed from the study prior to being randomized into an Arm.
Period: Overall Study
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks | Not Randomized to an Arm
Started | 53 | 54 | 27
Completed | 53 | 54 | 0
Not Completed | 0 | 0 | 27
Not completed — Determined to be ineligible | 0 | 0 | 16
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawn due to time of surgery being moved up. | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks | Not Randomized to an Arm | Total
Number analyzed (Participants) | 53 | 54 | 27 | 134
Age, Continuous [Median (Full Range); unit: years] | 57.91 [33.40 to 81.42] | 62.27 [32.22 to 86.86] | 65.46 [36.54 to 75.79] | 61.36 [32.22 to 86.86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 27 | 134
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 53 | 54 | 27 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 4 | 6 | 19
  White | 43 | 49 | 20 | 112
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 27 | 134

OUTCOME MEASURES:

1. Primary Outcome: Worst Pain as Measured by the Brief Pain Inventory (BPI) at 1 Year
Description: * The participant is asked to rate their pain by circling the one number that best describes their pain at its worst in the past week.
  * 0=no pain and 10 = pain as bad as they can imagine. The higher number indicates worse pain.
Time Frame: At 1 year
Population: Due to missing 1 year follow-up Brief Pain Inventories, all enrolled participants were not evaluable or included in this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks
Number analyzed (Participants) | 29 | 32
score on a scale | 0 [0 to 1] | 0 [0 to 0.8]
Statistical Analysis 1: Comparison: Preoperative PECS Blocks vs Placebo PECS Blocks; Test type: Superiority; p = 0.68, Kruskal-Wallis

2. Primary Outcome: Average Pain as Measured by the Brief Pain Inventory (BPI) at 1 Year
Description: * The participant is asked to rate their pain by circling the one number that best describes their pain on the average.
  * 0=no pain and 10 = pain as bad as they can imagine. The higher number indicates worse pain.
Time Frame: At 1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks
Number analyzed (Participants) | 29 | 32
score on a scale | 0 [0 to 0.2] | 0 [0 to 0.2]
Statistical Analysis 1: Comparison: Preoperative PECS Blocks vs Placebo PECS Blocks; Test type: Superiority; p = 0.67, Kruskal-Wallis

3. Primary Outcome: Interference as Measured by the Brief Pain Inventory (BPI) at 1 Year
Description: * The participant is asked circle the one number that describes how much, during the past week pain has interfered with general activity, mood, walking ability, normal work (includes both work outside the home and housework), relations with other people, sleep, and enjoyment of life.
  * 0=does not interference and 10 = completely interferes. The higher number indicates more interference from pain.
  * The scores for each subsection will be averaged.
Time Frame: At 1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks
Number analyzed (Participants) | 28 | 32
score on a scale | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Preoperative PECS Blocks vs Placebo PECS Blocks; Test type: Superiority; p = 0.53, Kruskal-Wallis

4. Secondary Outcome: Change in Quality of Life as Measured by the Veterans RAND12 Questionnaire Physical Health Summary Measure
Description: * The 12 items in the questionnaire correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The 12 items are summarized into two scores, a Physical Health Summary Measure (PCS) and a Mental Health Summary Measure (MCS).
  * The higher the score the better quality of life.
  * Scores are standardized to a mean of 50 with a range of -0.809-70.71.
Time Frame: At baseline and 1 year post-surgery
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks
Number analyzed (Participants) | 11 | 15
score on a scale | -3.1 [-18.0 to 1.9] | -0.8 [-10.3 to 7.8]
Statistical Analysis 1: Comparison: Preoperative PECS Blocks vs Placebo PECS Blocks; Test type: Superiority; p = 0.44, Kruskal-Wallis

5. Secondary Outcome: Change in Quality of Life as Measured by the Veterans RAND12 Questionnaire Mental Health Summary Measure
Description: * The 12 items in the questionnaire correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The 12 items are summarized into two scores, a Physical Health Summary Measure (PCS) and a Mental Health Summary Measure (MCS).
  * The higher the score the better quality of life.
  * Scores are standardized to a mean of 50 with a range of -1.465-77.09.
Time Frame: At baseline and 1 year post-surgery
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks
Number analyzed (Participants) | 11 | 15
score on a scale | 0 [-5.5 to 7.6] | 1.9 [-5.8 to 11.3]
Statistical Analysis 1: Comparison: Preoperative PECS Blocks vs Placebo PECS Blocks; Test type: Superiority; p = 0.88, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: -Adverse events will be tracked for 2 weeks after nerve block administration or patient discharge, whichever is later, up to 3 weeks. Most patients will be discharged within 24 hours. Adverse events thought to be at least possibly related to surgery will not be collected. -All-cause mortality was collected from day of surgery through completion of follow-up, up to 1 year. The one mortality occurred during follow-up and attribution to the PECS block was deemed as unrelated.
Description: Participants in the Not Randomized Arm were not assess for Serious and Other Adverse Events as they did not receive any study treatment or placebo.
Groups:
- Not Randomized to an Arm: -Participants were removed from the study prior to being randomized into an Arm and did not receive any treatment on the study.
Arm/Group | Preoperative PECS Blocks | Placebo PECS Blocks | Not Randomized to an Arm
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/54 | 1/27
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/0
Other Adverse Events (participants affected / at risk) | 5/53 | 0/54 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative PECS Blocks (N=53) | Placebo PECS Blocks (N=54) | Not Randomized to an Arm (N=0)
Hematoma (Vascular disorders) | 2 | 0 | NA
Swelling (General disorders) | 1 | 0 | NA
Seroma (Injury, poisoning and procedural complications) | 2 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03084536/Prot_SAP_000.pdf